CLINICAL TRIAL: NCT00889057
Title: Phase II, Open Label, Non-randomized Study of Second or Third Line Treatment With Sorafenib (BAY 43-9006) in Patients Affected by Relapsed High-grade Osteosarcoma.
Brief Title: Sorafenib in Relapsed High Grade Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Responsible Party: Principal Investigator, Prof. Massimo Aglietta, Professor, Italian Sarcoma Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGosteo-BAY; EudraCT Number: 2007-004396-19
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma; sorafenib; target therapy
MeSH Terms: conditions — Osteosarcoma | interventions — Sorafenib

ARMS (1):
- sorafenib (Experimental)
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — 400 mg bid until progression or inacceptable toxicity

SUMMARY:
Aim of this exploratory phase II study is to assess the clinical activity of sorafenib as single agent, in terms of percentage of patients with high grade advanced osteosarcoma free from progression following 4 months of therapy

ELIGIBILITY:
Inclusion Criteria:

* histologically documented and not surgically resectable or metastatic high-grade osteosarcoma which progressed after first or second line treatments for relapsing disease.
* measurable disease as defined by having at least one lesion that can be accurately measured by means of CT or MRI.
* ECOG PS of 0, 1 and an estimated life expectancy of at least 3 months. ECOG P.S. 2 is acceptable provided that it depends solely on orthopedic problems
* Age ≥15 years.
* Adequate bone marrow, liver and renal function
* Written informed consent

Exclusion Criteria:

* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Coexisting malignancies, except for basal or epithelial cell carcinoma of the skin or other solid tumors curatively treated with no evidence of disease for ≥3 years.
* History of cardiac disease: congestive heart failure >NYHA class 2; active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
* History of HIV infection or chronic hepatitis B or C.
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
* Patients with seizure disorders requiring medication (such as steroids or anti-epileptics)
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and two weeks after the completion of trial.
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Patients unable to swallow oral medications

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Tumor assessment through radiologic evaluation. | every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Aglietta, MD, Study Chair — I.R.C.C - FPO Candiolo; Giovanni Grignani, MD, Principal Investigator — I.R.C.C. - FPO Candiolo
Locations (4):
- Italy (4):
  - Istituti Ortopedici Rizzoli - Unit of Chemotherapy of Muscoloskeletal Tumors, Bologna, Bologna
  - Istituto Nazionale Tumori - Unit of Medical Oncology, Milan, Milano
  - I.R.C.C. - Unit of Medical Oncology, Candiolo, Torino
  - Ospedale Infantile Regina Margherita - Unit of Paediatric Oncoematology, Torino, Torino